CLINICAL TRIAL: NCT01157910
Title: An Epidemiological and Bacteriological Assessment of Middle Ear Fluid in Children Undergoing Ventilation Tube Placement Surgery
Brief Title: Bacterial Assessment of Middle Ear Fluid in Children Undergoing Ventilation Tube Placement Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Dr. Shimon Schreiber, Hillel Yaffe Hospital, Department of Ear Nose And Throat
Other Study IDs: 36-2009
Record Dates: First submitted 2010-07-04; First posted 2010-07-07 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Chronic Otitis Media; Age Determined Bacteria
Keywords: Ear infection; Chronic
MeSH Terms: conditions — Otitis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Children with chronic otitis media have more resistant bacteria that require surgical intervention to eradicate the infections. The study will evaluate the dominant bacteria and their sensitivities to antibiotics. The information will assist in better treatment plans for children with chronic infections.

The data will also assess the changing patterns in the bacteria colonizing middle ear fluid.

DETAILED DESCRIPTION:
ibid.

ELIGIBILITY:
Inclusion Criteria:

* All children with chronic ear infections scheduled for surgical interventions

Exclusion Criteria:

* Children who have undergone prior mastoid surgery, or children with oncologic treatments.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children suffering from chronic otitis media who are scheduled for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-11 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe MC,, Hadera, Israel